CLINICAL TRIAL: NCT07115160
Title: The Leksand Hockey Trial on Grip Strength
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dalarna County Council, Sweden (Other)
Responsible Party: Principal Investigator, Daniel Muder, MD, PhD, Dalarna County Council, Sweden
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2024-08560-01
Record Dates: First submitted 2025-06-20; First posted 2025-08-11 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-10

CONDITIONS: Grip Strength; Performance; Injuries
Keywords: grip strength; ice hockey; injury; professional; performance; game score; sports science; strength training; athletes
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Intervention Model Description: In the second phase of the study, a standardized grip strength training program will be implemented as the primary intervention. This program is designed to improve grip strength in professional hockey players over a defined period (details in Appendix D). All participants who completed Phase 1 will undergo this intervention.
  The training program includes specific exercises targeting the forearm flexors and extensors, wrist stability, and hand grip endurance. Typical exercises may involve hand grippers, wrist rollers, towel wringing, plate pinches, and resisted squeezing movements using elastic bands or putty. Training frequency, intensity, duration, and progression will be standardized and supervised to ensure consistency across participants.
  After completion of the training period, grip strength will be re-measured using the same HAKIR protocol and dynamometer. Performance metrics-game score, shots on goal, and shooting precision-will also be collected for the five games following
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Grip Strength Training (Experimental): In the second phase of the study, a standardized grip strength training program will be implemented as the primary intervention. This program is designed to improve grip strength in professional hockey players over a defined period (details in Appendix D). All participants who completed Phase 1 will undergo this intervention.
  The training program includes specific exercises targeting the forearm flexors and extensors, wrist stability, and hand grip endurance. Typical exercises may involve hand grippers, wrist rollers, towel wringing, plate pinches, and resisted squeezing movements using elastic bands or putty. Training frequency, intensity, duration, and progression will be standardized and supervised to ensure consistency across participants.
  After completion of the training period, grip strength will be re-measured using the same HAKIR protocol and dynamometer. Performance metrics-game score, shots on goal, and shooting precision-will also be collected for the five games following
  Interventions: Other: Training following a predefined protocol.

INTERVENTIONS:
Other: Training following a predefined protocol. — Training following a predefined protocol.

SUMMARY:
This project, titled The Leksand Hockey Trial on Grip Strength, investigates whether grip strength is related to performance in professional hockey players. Grip strength is already known to reflect general health and muscle function, and it plays a key role in ice hockey, where players rely on strong hands and forearms for stick handling, shooting, and physical challenges on the ice. Despite this, no clinical study has yet explored whether stronger grip strength leads to better on-ice performance. In this pilot study, we will first examine if there is a correlation between grip strength and key performance indicators such as game score (a combined measure of offensive and defensive contribution), number of shots on goal, and shooting precision. Grip strength will be measured using a standardized protocol and professional players from SHL, SDHL, and HockeyAllsvenskan will be included. Performance data will be collected before and after the grip strength assessment. Additionally, injuries sustained during the study period will be recorded and monitored as an outcome measure. We will investigate whether there is any correlation between grip strength and injury incidence to assess if stronger grip strength may influence injury risk or resilience in professional hockey players. In the second part of the study, players will follow a grip-strength training program to determine whether improvements in grip strength lead to better performance. If a link is found, grip strength could be used as a simple and reliable proxy for player performance and may justify the inclusion of specific grip training in professional hockey conditioning programs. This study aims to fill a knowledge gap in elite sports science and could help optimize training and evaluation methods in professional ice hockey.

DETAILED DESCRIPTION:
This study, titled The Leksand Hockey Trial on Grip Strength, aims to explore the relationship between grip strength (GS) and athletic performance in professional ice hockey players. Grip strength is a well-established biomarker for general muscle function, physical capability, and even long-term health outcomes. It is commonly used in sports medicine, rehabilitation, and performance diagnostics due to its simplicity, reliability, and cost-effectiveness. In ice hockey, grip strength plays a particularly critical role given the physical demands of stickhandling, shooting, passing, puck control, and body contact situations.

Despite its relevance, the correlation between grip strength and actual game performance in elite hockey players has not been systematically studied. This project addresses two primary research questions: (1) Does grip strength correlate with performance in professional hockey players? and (2) Does improved grip strength result in measurable performance improvements?

The study will be conducted in two phases. In Phase 1, we will recruit approximately 40 professional male and female hockey players from the Swedish Hockey League (SHL), Swedish Women's Hockey League (SDHL), and HockeyAllsvenskan. Each participant will undergo grip strength testing using the standardized HAKIR protocol with a Jamar dynamometer. Three alternating trials per hand will be recorded, and the average grip strength (in kilograms) will be calculated. Simultaneously, player performance will be assessed based on three key metrics:

Game Score: A composite metric capturing offensive and defensive contributions, adjusted for even-strength playing time (adapted from existing SHL models).

Shots on Goal: Total number of shots per game.

Shooting Precision: Ratio of goals to total shots taken.

Injuries sustained during the season

Each of these metrics will be collected for the five games preceding and following grip strength measurement. Statistical analyses will include Pearson correlation, t-tests, chi-square tests, and non-parametric alternatives where appropriate. Estimates will be presented with 95% confidence intervals, and p-values < 0.05 will be considered statistically significant. As a pilot study, no formal power calculation will be performed initially, but variance estimates will be used to plan a larger future trial.

Additionally, injuries sustained during the study period will be recorded and monitored as an outcome measure. We will investigate whether there is any correlation between grip strength and injury incidence to assess if stronger grip strength may influence injury risk or resilience in professional hockey players.

In Phase 2, participants will engage in a standardized grip-strength training program over a defined period (see Appendix D). Post-intervention grip strength and performance metrics will be reassessed using the same methods to determine whether an increase in grip strength is associated with performance improvement.

Inclusion criteria include:

Active rostered player in SHL, SDHL, or HockeyAllsvenskan

No current hand or wrist injury

Exclusion criteria:

Not currently signed in the aforementioned leagues

Current injury to the hand or wrist that impairs testing

This project addresses a notable knowledge gap in elite performance research. If grip strength is shown to correlate with or enhance performance, it could be used as a proxy marker in sports performance evaluations and as a justification for implementing targeted grip-strength training in professional hockey conditioning programs. The findings may contribute to improved training strategies, rehabilitation protocols, and performance monitoring in elite ice hockey.

ELIGIBILITY:
Inclusion Criteria:

* Professional hockey player signed in the SHL/SDHL/Hockey Allsvenskan
* No current hand injury

Exclusion Criteria:

* Not signed in the SHL/SDHL/Hockey Allsvenskan
* Current hand injury

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-11-05 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Game Score | Calculated for each player at baseline and at follow-up, which will occur no earlier than 10 weeks and no later than 24 weeks.
  The Game Score used in this study is calculated as follows:
  Game Score = Offensive Game Score + Defensive Game Score
  Each component is defined below:
  Offense:
  Individual Contributions:
  * Goal: 0.75
  * First assist: 0.7
  * Second assist: 0.55
  * Expected goals (xG): 0.5
  On-ice Contributions (team performance with the player on the ice):
  * Goals for: 0.625 (for forwards), 0.425 (for defensemen)
  * Shots attempted for: 0.625 (for forwards), 1.7 (for defensemen)
  Defense:
  Individual Contributions:
  • Penalty minutes: 0.15
  On-ice Contributions (team performance with the player on the ice):
  * Goals against: 0.4375 (for forwards), 0.575 (for defensemen)
  * Shots attempted against: 1.75 (for forwards), 2.3 (for defensemen) Each component is adjusted based on the player's minutes played in each game and is measured in goals above average.

SECONDARY OUTCOMES:
Shots on goal/game | Calculated for each player at baseline and at follow-up, which will occur no earlier than 10 weeks and no later than 24 weeks.
  Number of shots on goal/game
Shooting prescision | Calculated for each player at baseline and at follow-up, which will occur no earlier than 10 weeks and no later than 24 weeks.
  To measure shooting accuracy by counting successful shots on two designated target areas in the goal.
  Equipment and Setup:
  Player Equipment: Standard training gear used in regular practice.
  Puck: Standard SHL/SDHL hockey puck.
  Goal: Standard SHL/SDHL goal.
  Targets: Two targets at:
  Upper left corner (1)
  Upper right corner (2) Each ~13 cm (5 inches) diameter.
  Distance: Player positioned 4-5 meters (13-16 feet) directly in front of the goal.
  Procedure:
  Pre-Test Preparation:
  Conducted during or immediately after a regular training session.
  Players complete standard warm-up.
  Shooting Protocol:
  Each player completes 15 shots per target, alternating every 5 shots between the upper left and upper right corners.
  Total of 30 shots per player.
  Observers record hit/miss on a simple tally sheet.
Injuries | From the start of the 2025/26 season on September 13th until the end of the season, defined by the date of the final playoff game.
  Injuries reported during the season. Regarding type of injury and missed ice time due to the injury.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Muder, MD, PhD, Principal Investigator — Centre for Clinical Research Dalarna, Uppsala University, Sweden
Locations (1):
- Leksands IF, Leksand, Region Dalarna, Sweden

IPD SHARING:
Plan to Share IPD: Yes
Any data shared with colleagues or collaborating researchers will be fully anonymized or pseudonymized to protect participant privacy in accordance with GDPR regulations. Data transfers will occur under strict confidentiality agreements, and all parties will adhere to applicable data protection laws to ensure the security and privacy of personal information. We will act in accordance with the ethical approval granted by the Swedish Ethical Review Authority (EPM) and comply with all relevant local policies regarding data protection.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: From the publication of the protocol and for 10 years thereafter.
Access Criteria: Access to individual participant data is typically restricted to authorized researchers involved in the study or approved collaborators under strict confidentiality and data protection agreements.

REFERENCES:
- [Background] Jiang R, Westwater ML, Noble S, Rosenblatt M, Dai W, Qi S, Sui J, Calhoun VD, Scheinost D. Associations between grip strength, brain structure, and mental health in > 40,000 participants from the UK Biobank. BMC Med. 2022 Sep 9;20(1):286. doi: 10.1186/s12916-022-02490-2. PMID 36076200
- [Background] Toong T, Wilson KE, Urban K, Paniccia M, Hunt AW, Keightley M, Reed N. Grip Strength in Youth Ice Hockey Players: Normative Values and Predictors of Performance. J Strength Cond Res. 2018 Dec;32(12):3494-3502. doi: 10.1519/JSC.0000000000002815. PMID 30216250
- [Background] Tavares Junior AC, Silva HS, Penedo T, do Amaral Rocha LGS, da Silva AS, Venditti Junior R, Dos-Santos JW. Correlation of the Handgrip Strength and Body Composition Parameters in Young Judokas. Int J Environ Res Public Health. 2023 Feb 2;20(3):2707. doi: 10.3390/ijerph20032707. PMID 36768073
- [Background] Trivic T, Eliseev S, Tabakov S, Raonic V, Casals C, Jahic D, Jaksic D, Drid P. Somatotypes and hand-grip strength analysis of elite cadet sambo athletes. Medicine (Baltimore). 2020 Jan;99(3):e18819. doi: 10.1097/MD.0000000000018819. PMID 32011492
- [Background] Roberts HC, Denison HJ, Martin HJ, Patel HP, Syddall H, Cooper C, Sayer AA. A review of the measurement of grip strength in clinical and epidemiological studies: towards a standardised approach. Age Ageing. 2011 Jul;40(4):423-9. doi: 10.1093/ageing/afr051. Epub 2011 May 30. PMID 21624928
- [Background] Ewing Fess, E. Clinical Assessment Recommendations. Michigan: In Casanova, J. S. (Ed.),American Society of Hand Therapists.; pp. 41-45). (2d edition; vol. 1992).
- See also: Introduction to game score. — https://hockey-graphs.com/2016/07/13/measuring-single-game-productivity-an-introduction-to-game-score/
- See also: Information on game score. — https://en.wikipedia.org/w/index.php?title=Game_score&oldid=1246967719